CLINICAL TRIAL: NCT03961113
Title: Pilot Study of the Impact of Giant Cell Arteritis and Its Treatment on the Autonomy of the Elderly in the First Year of Care
Acronym: EPACAPA
Status: Terminated | Type: Observational
Why Stopped: inadequate recruitment
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0008 (EPACAPA)
Record Dates: First submitted 2019-05-17; First posted 2019-05-23 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Giant Cell Arteritis in Dependency of Elderly
Keywords: Giant Cell Arteritis; Dependency; Elderly
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessment by questionnaire
  Interventions: Other: Assessment by questionnaire

INTERVENTIONS:
Other: Assessment by questionnaire — At diagnosis a gerontological evaluation will be carried out including the following tests: ADL, iADL, MNA, SF 36, SPPB, FRIED criteria and GDS. The set of scales and scores of the procedure is commonly used in geriatrics to assess the fragility of the patient.
  A monthly telephone reassessment conducted by an ARC will collect ADL and iADL from the first month to the eleventh month. The end-of-study consultation will be conducted by a geriatrician at the 12th month and will include the following tests: ADL, iADL, MNA, SF 36, the SPPB, the criteria of FRIED and the GDS

SUMMARY:
Giant cell arteritis is the leading cause of vasculitis in the elderly. No work evaluates its impact on autonomy. At the diagnosis a gerontological evaluation will be carried out including the scores ADL, iADL, MNA, SF 36, SPPB, FRIED and GDS. A monthly telephone reassessment will collect ADL and iADL. The end-of-study consultation at M12, conducted by a geriatrician, will have the same scores as at M0. This will make it possible to evaluate the difference in the functional autonomy score between M0 and M12 in the elderly with ACG.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65 years with at least 2 comorbidities * present, or age greater than or equal to 75 years
* Diagnosis of ACG meeting the diagnostic criteria of ACG 1990 ACR

  * comorbidity = chronic pathology

Exclusion Criteria:

* Neoplastic pathology under treatment
* Brain pathology with motor disability
* Dementia at a severe stage (MMS <22/30)
* Unable to answer the phone
* Participation in a therapeutic clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patient with giant cell arteritis
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Activities of Daily Living (ADL) | Month 12
  Compare score between Month 0 and Month 12. The scale is evaluated from 0 (dependence) to 6 (autonomy).

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) | Month 11
  Compare the evolution every month at M0 and every month up to Month 11 The scale is evaluated from 0 (dependence) to 6 (autonomy).

OTHER OUTCOMES:
Instrumental Activities of Daily Living (iADL) | Month 12
  Compare the evolution every month at Month 0 and every month up to Month 12 The scale is evaluated from 0 (dependence) to 8 (autonomy).
Mini Nutritional Assessment (MNA) | Month 12
  Compare score between Month 0 and Month 12 The scale is evaluated from 0 (poor nutritional status) to 30 (correct)
The Short Form Health Survey (SF-36) : Physical score | Month 12
  Compare score between Month 0 and Month 12 The scale is evaluated from 13,6 (poor physical condition) to 61.9 (good physical condition)
The Short Form Health Survey (SF-36) : Psychic score | Month 12
  Compare score between Month 0 and Month 12 The scale is evaluated from 15.6 (poor psychic condition) to 70 (good physical condition)
Short Physical Performans Battery (SPPB) | Month 12
  compare score between Month 0 and Month 12 The scale is evaluated from 0 (poor performance) to 12 (high performance)
fragility criteria questionnaire (Fried) | Month 12
  compare score between Month 0 and Month 12 The scale is evaluated from 0 (robust) to 5 (fragile)
Geriatric Depression Scale (GDS) | Month 12
  compare score between Month 0 and Month 12 The scale is evaluated from 0 (normal) to 30 (severe depression)
The cumulative dose of corticosteroids and autonony loss | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France